CLINICAL TRIAL: NCT04115241
Title: Activity Levels in Bone Marrow Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Michael Tomasson (Other)
Responsible Party: Sponsor-Investigator, Michael Tomasson, Professor Internal Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202208637-B
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bone Marrow Transplant
Keywords: leukemia; multiple myeloma; myelodysplastic syndrome; stem cell transplant
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Actigraph — Actigraphs are non-invasive, wearable devices that measure activity levels using an accelerometer
Other: Grip strength test — The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles

SUMMARY:
Participants in this study will be receiving a bone marrow transplant. This study is designed to evaluate correlations between activity levels and length of stay, quality of life, and hand grip strength.

DETAILED DESCRIPTION:
Participants in this study will be receiving a bone marrow transplant. Participants will be given actigraphs to wear around their waists starting 3 weeks prior to bone marrow transplants until they are discharged from the hospital. Participants will be asked to complete quality of life questionnaires and hand grip tests at three separate time points during their hospitalizations. All data gathered from these activities will be compared with patients' activity levels gathered from the actigraphs both before and during the hospitalization. This study is designed to determine the relationship between activity levels and length of stay, quality of life, and hand grip strength.

ELIGIBILITY:
Patients who will be receiving a bone marrow transplant are eligible for this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be receiving a bone marrow transplant
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2030-05-23 (Estimated); Study Completion 2030-05-23 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation between activity levels and length of stay in hospital | From study intitiation for up to 5 years
  Participants will be given actigraphs to wear around their waists starting 3 weeks prior to bone marrow transplants until they are discharged from the hospital. Activity prior to and during hospitalization will be correlated with length of stay.
To determine the correlation between activity levels and quality of life | From study intitiation for up to 5 years
  Participants will be given actigraphs to wear around their waists starting 3 weeks prior to bone marrow transplants until they are discharged from the hospital. They will be provided with quality of life questionnaires at three time points during hospitalization. Activity prior to and during hospitalization will be correlated with quality of life
To determine the correlation between activity levels and hand grip strength | From study intitiation for up to 5 years
  Participants will be given actigraphs to wear around their waists starting 3 weeks prior to bone marrow transplants until they are discharged from the hospital. Hand grip strength will be measured at three time points during hospitalization. Activity prior to and during hospitalization will be correlated with hand grip strength.

SECONDARY OUTCOMES:
To determine barriers to activity for patients recovering from bone marrow transplantation and design an intervention to increase activity levels in patients post-transplantation | From study intitiation for up to 5 years
  Barriers to physical activity will be determined using a validated questionnaire at three time points during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tomasson, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No